CLINICAL TRIAL: NCT02954640
Title: Evaluation of the Efficacy of the Sequencing Method by Gene-panel, Compared to the Reference Sanger Method, on Patients With Primary Immuno-deficiencies, and Who Need a Genetic Diagnosis.
Brief Title: Evaluation of the Efficacy of the Sequencing Method by Gene-panel
Acronym: Génétique-DIH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Imagine Institute (Other)
Collaborators: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IMIS2015-02
Record Dates: First submitted 2016-11-02; First posted 2016-11-03 (Estimated); Last update posted 2018-03-15 (Actual); Status verified 2018-03

CONDITIONS: Primary Immuno-Deficiencies
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Patient with PID (Other): For patient with clinical diagnosis of PID, an additional blood sampling will be taken.
  The genetic diagnosis will be done via the method of gene-panel in the frame of the study.
  A genetic confirmation will, in any case, be done via the reference method (Sanger), in order to establish a final diagnosis for these patients.
  Interventions: Biological: Blood sampling

INTERVENTIONS:
Biological: Blood sampling — Additional blood sampling for the realization of the test on the gene panel

SUMMARY:
In order to accelerate the identification of genes responsibles of PID, and to improve the diagnosis of PID, the research team would like to validate a rapid and targeted method of high-throughput sequencing, on 301 genes, known to be involved in PID.

DETAILED DESCRIPTION:
The Primary Immuno-Deficiencies (PID) are a set of rare diseases (estimated incidence of 1/5000). Today, more than 320 PID are described, and for 301 of them, the genetic cause has been identified, which underlines the huge diversity of all PID.

The genetic diagnosis of PID is very important for the comprehension of PID physiopathology, their treatment and the genetic patient information.

The characterisation of the clinical and immunological phenotype of patients allowed to identify a known morbid gene in 30% of cases, but for other patients, the genetic cause remains unknown, due to, inter alia, the lack of efficient tools for genetic exploration.

In this context, each year, around 600 French and foreign patients are explored at the Necker hospital CEDI (Center for Immuno-Deficiencies Explorations), for whom are identified, in 30% of cases, a known genetic cause.

Their treatment and the diagnosis of these patients is slow, partially because these studies are dependants of research fundings. In addition, in the current practice, the investigators sometimes discover incidental findings via the non-targeted high throughput genetic analyzes.

The aim of the gene-panel is to improve the diagnosis procedures of these known diseases, by generalizing a rapid and targeted method of sequencing, on 301 genes, known to be involved in PID.

ELIGIBILITY:
Inclusion Criteria:

* Patient who need a genetic diagnosis of PID done at Necker's CEDI (Center for Immuno-Deficiencies Explorations), in the frame of an initial causal mutation identification
* Patient having signed an informed consent form (or parents for minor patients)
* Patient affiliated to National Health Care Insurance

Exclusion Criteria:

* Patient refusing to participate
* Patient under legal guardianship
* Patient that can't fulfill the study requirements, for any geographic, social or psychic reason

Max Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2016-02; Primary Completion 2017-09-08 (Actual); Study Completion 2017-09-08 (Actual)

PRIMARY OUTCOMES:
Comparison of the 2 sequencing methods | 2 years
  Assess the efficacy of the identification of the genetic cause of PID, via the high throughput gene panel sequencing method, compared to the reference Sanger method, on patients with no identified mutation after analyzes done by available technics on hospital laboratories.

CONTACTS AND LOCATIONS:
Overall Officials: Alain Fischer, Study Chair — Imagine Institute; Alexandre Alcais, Study Chair — Imagine Institute
Locations (1):
- Necker - Enfants Malades hospital, Paris, France

IPD SHARING:
Plan to Share IPD: No